CLINICAL TRIAL: NCT00081068
Title: Phase II Study of Campath-1H in Lymphoplasmacytic Lymphoma (Waldenstrom's Macroglobulinemia)
Brief Title: Alemtuzumab in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000358811; UCLA-0309058
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Alemtuzumab

INTERVENTIONS:
Biological: alemtuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: This phase II trial is studying how well alemtuzumab works in treating patients with Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response in patients with Waldenstrom's macroglobulinemia treated with alemtuzumab.
* Determine the time to treatment failure in patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive alemtuzumab IV over 2 hours on days 1, 3, and 5 of weeks 1-6 (course 1) in the absence of disease progression or unacceptable toxicity. Patients with a complete response undergo observation. Patients with stable disease or a minor or partial response receive an additional course of alemtuzumab, administered as in course 1, on weeks 7-12.

Patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 13-27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Waldenstrom's macroglobulinemia (lymphoplasmacytic lymphoma)

  * Immunoglobulin (Ig) M, IgG, and IgA paraprotein
  * Measurable monoclonal paraprotein
* Failed at least 1 prior first-line therapy (alkylator agent, nucleoside analogue, or rituximab)
* CD52-positive tumor determined by either bone marrow immunohistochemistry or flow cytometry

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Absolute neutrophil count ≥ 500/mm^3
* Platelet count ≥ 25,000/mm^3

Hepatic

* SGOT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN

Renal

* Creatinine ≤ 2.5 mg/dL (> 2.5 mg/dL allowed if due to disease)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception during and for 6 months after study participation
* No serious comorbid disease
* No uncontrolled bacterial, fungal, or viral infection
* No other active malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior alemtuzumab
* More than 3 months since other prior monoclonal antibody therapy

Chemotherapy

* See Disease Characteristics
* More than 21 days since prior chemotherapy

Endocrine therapy

* More than 21 days since prior steroid therapy

Radiotherapy

* More than 21 days since prior radiotherapy

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-01

PRIMARY OUTCOMES:
Objective response
Time to treatment failure
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gansert, MD, PhD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (15):
- United States (10):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Rocky Mountain Cancer Centers - Denver Midtown, Denver, Colorado
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia
- Canada (2):
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Centre Hospitalier Lens, Lens, France
- Saint Bartholomew's Hospital, London, England, United Kingdom